CLINICAL TRIAL: NCT05860725
Title: Appalachian Voices for Health - Feasibility Trial of a Multi-level Media Production and Social Marketing Campaign to Reduce HPV Vaccine Hesitancy
Brief Title: Feasibility Trial of a Multi-level Media Production and Social Marketing Campaign to Reduce HPV Vaccine Hesitancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Kathleen Porter, Phd, RD, Assistant Professor, University of Virginia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SBS-5519
Record Dates: First submitted 2023-02-28; First posted 2023-05-16 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Human Papillomavirus Infection; Vaccination Hesitancy
MeSH Terms: conditions — Papillomavirus Infections; Vaccination Hesitancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PSA Development (Phase 1) (Experimental)
  Interventions: Behavioral: PSA Development
- Social Marketing Campaign (Phase 2) (Experimental)
  Interventions: Behavioral: HPV vaccination focused social marketing campaign
- Organizational Stakeholders (No Intervention): Organizational stakeholders from organizations involved in Phase 1 and 2 will take part in a focus group after their respective phases have been completed to learn more about their experience.

INTERVENTIONS:
Behavioral: PSA Development — Health sciences students from a regional community college in Appalachian Virginia will be asked to to develop and submit a public service announcement (PSA) and to watch virtual training webinars that support the development of the PSAs. They will also be asked to complete surveys at three time points: before the PSA contest starts, after the PSA contest ends, and upon submitting a PSA.
  Arms: PSA Development (Phase 1)
Behavioral: HPV vaccination focused social marketing campaign — Community members who use a regional health services focused non-profits rideshare buses and/or view their social media pages will be exposed to a 12-week social marketing campaign that uses PSAs developed in Phase 1. Community members will also complete surveys at three time points: before the start of the social marketing campaign, during the social marketing campaign, and after the social marketing campaign.
  Arms: Social Marketing Campaign (Phase 2)

SUMMARY:
Since 2019, the HPV working group of the University of Virginia Cancer Center's Southwest Virginia Community Advisory Board has developed and executed strategies to increase regional HPV vaccination rates. Members collaboratively developed Appalachian Voices for Health, a multi-level media production and social marketing intervention. This novel intervention builds on the past efforts of the working group and the engaged organizations; takes into account the impact of vaccine hesitancy on HPV vaccination uptake; and incorporates best practices. Through the intervention, Nursing and Dental Assistant students from Mountain Empire Community College will develop PSAs after receiving training about HPV vaccination and health communication. These PSAs will be used in a social marketing campaign executed through a regional transportation system managed by Mountain Empire Older Citizens. Specifically, the trial's aims are three-fold: assess the intervention's impact on community members' and students' HPV vaccine hesitancy (Aim 1) and perceptions and actions related to HPV vaccination (Aim 2) and evaluate other feasibility indicators at the community-, student-, organizational-, and process levels (Aim 3). The research team will use a concurrent mix-methods approach to assess feasibility indicators. Aims will be assessed using surveys, focus groups, meeting minutes, and implementation records. Data will be analyzed using descriptive and inferential statistics and content coding. Determination of the intervention's feasibility will consider the achievement benchmarks for feasibility indicators individually and collectively. Data will be used to inform refinement and future testing of Appalachian Voices for Health.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* enrolled as a student in one of the regional community college's health sciences programs (Phase 1 only)
* ride the regional health services focused non-profit's rideshare buses or view their social media during one or more of the three survey periods (Phase 2 only)
* work for either the regional community college or non-profit AND were involved in supporting the execution of the study components within their organization.

Exclusion Criteria:

* Under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Vaccination hesitancy scale modified for the HPV vaccine (VHS-HPV) | Change in community members' self-reported VHS-HPV score pre-post intervention (14 week period / Phase 2)
  validated instrument; 9 items on a response scale of 1-5 (strongly disagree to strongly agree) with higher scores indicating greater hesitancy
Vaccination hesitancy scale modified for the HPV vaccine (VHS-HPV) | Change in Health Sciences students' self-reported VHS-HPV score pre-post intervention (6 week period / Phase 1)
  validated instrument; 9 items on a response scale of 1-5 (strongly disagree to strongly agree) with higher scores indicating greater hesitancy

SECONDARY OUTCOMES:
Vaccination hesitancy scale (VHS) | Change in community members' self-reported VHS score pre-post intervention (14 week period / Phase 2)
  validated instrument; 10 items on a response scale of 1-5 (strongly disagree to strongly agree) with higher scores indicating greater hesitancy
Vaccination hesitancy scale (VHS) | Change in Health Science students' self-reported VHS score pre-post intervention (6 week period / Phase 1)
  validated instrument; 10 items on a response scale of 1-5 (strongly disagree to strongly agree) with higher scores indicating greater hesitancy

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No